CLINICAL TRIAL: NCT06269471
Title: Prevalence and Impact of Chronic Ankle Instability in Trailers : an Epidemiological Study on French Trails
Brief Title: On the ICC's Path: a Prevalence Study
Acronym: SSICC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02039-36
Record Dates: First submitted 2023-12-04; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Chronic Ankle Instability
Keywords: Chronic Ankle Instability; Trail Running; Ultra Trail Running; Ankle Sprain; Prevalence
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trailers: Group of major trail runners who have already taken part in at least one trail running competition in their lives.

SUMMARY:
The number of trailers is growing all the time, and TRu seems to be a risky activity for the ankle joint. Ankle sprains can lead to significant health consequences, as in the case of chronic ankle instability.

However, there are no studies informing of the prevalence of chronic ankle instability in trail running. The aim of this study is therefore to take stock of chronic ankle instability in trail running in France.

DETAILED DESCRIPTION:
Trail Running Trail running (TRu) is a running sport that abounds in creativity in the composition of its courses. It is the most popular sport in off-road running. The International Trail Running Association (ITRA), TRu's international governing body since 2013, with the International Association of Ultrarunners (IAU), manages and develops ultra-distance races under the patronage of the International Association of Athletics Federations (IAAF). They defines TRu as running in a natural environment including mountains, deserts, forests, coastal areas, jungles or rainforests, grassy or arid plains over a variety of different terrains with a minimum of paved or asphalt roads (not exceeding 20 to 25% of the total course). TRu can be practiced in competitions open to all, in semi-self-sufficiency or in self-sufficiency. The latter takes place with respect for sporting ethics, fairness, solidarity and the environment. This sport differs from Ultra Trail Running in terms of distance. Indeed, any race longer than a marathon, i.e. 42.195km, qualifies as an Ultra. On the other hand, there is no difference or restriction as to the altitude difference covered.

According to the Fédération Française d'Athlétisme (FFA), there are now over 800,000 TRu enthusiasts in France and 20 million worldwide. For more than ten years, this outdoor sport, whose popularity grew with the Covid-19 pandemic, has been growing at an annual rate of around 12% worldwide. The year 2022, for example, saw a massive expansion, with more Trail Running events than road races recorded in France for the first time (3035 versus 2706). This represents an average of almost 418 events scheduled every weekend for TRu enthusiasts.

Ankle sprains Among the most common sports pathologies, lateral ankle sprains are the most common, well ahead of muscle injuries and tendinopathies. In 2015 in France, there were nearly 6,000 cases of ankle sprains every day, corresponding to more than 1.2 million euros in just 24 hours. In other words, 70% of the population has already suffered a sprain in the course of their life. These figures reflect a real public health problem.

Ankle sprain is described as a "condition resulting from distortion beyond physiological limits during forced, abrupt movement of the hindfoot without permanent bony displacement". Four different types of ankle sprains are usually reported, including lateral talocrural sprain (the most common), medial talocrural sprain (extremely rare), subtalar sprain and anterior sprain. In 95% of cases, the injury involves the lateral collateral ligament plane. The patho-mechanics of this injury correspond to a sequence of forced inversion associated with pure varus, internal rotation, forced plantar flexion, and forced eversion.

Chronic ankle instability Ankle sprains have the highest recurrence rate of all lower-limb injuries, and in 40% of cases develop into chronic instability. Following a first episode, 70% of people will suffer a recurrence. In fact, this risk doubles the following year. Poor management of ankle sprains can have significant consequences for the joint and its function.

According to the new model updated by Hertel, chronic ankle instability (CAI) is defined by 8 elements. These include the sprain and associated primary tissue damage, environmental factors, personal factors, patho-mechanical impairments, perceptual and sensory impairments, behavioral and motor impairments, the interactions between each element and the spectrum of clinical outcomes. A patient with CHF, however, does not systematically possess each of these impairments.

Copers patients The mere presence of an ankle sprain does not determine the evolution of this injury into chronic instability. Indeed, so-called "Copers" patients have suffered a lateral ankle sprain but have not developed a sensation of instability or sprain recurrence after 12 months. The explanations for this recovery are multiple and specific to each patient.

The Cumberland Ankle Instability Tool Several diagnostic tools can be used to assess CCI. The International Ankle Consortium recommends the use of the Cumberland Ankle Instability Tool as a validation questionnaire specific to chronic ankle instability. The CAIT consists of 9 items in a 30-point format to measure the severity of functional ankle instability (FAI). This validated self-questionnaire distinguishes between people with CAI and those without (p<0.001), with a threshold score ≤ 23 points for the French version and ≤ 25 for the English version. Significant correlations were observed between the CAIT, the LEFS and the VAS, other validated questionnaires, in addition to excellent test-retest reliability. The translation of this self-questionnaire involves different threshold scores (≤23 and ≤25) respectively validated.

Data on ankle sprain and TRu PubMed lists over 2,234 results for the keyword "ankle chronic instability". A search for the keywords "ankle chronic instability" AND "sport", reveals 503 corresponding studies, i.e. 4 times fewer. A search of "ankle chronic instability" AND "running", reveals almost 48 results. Despite this, the new combination of "ankle chronic instability" AND "trail running" yields no published studies. The terms "outdoor", "mountain", "ultra trail running" or "hiking" also produced no results.

Given the increase in practice and the lack of data, further research is paramount knowledge about chronic ankle instability in TRu. There are good reasons to believe that ankle injuries are frequent in this sport and that they can have significant consequences.

Objectives As a first step, investigators will study the prevalence of CCI among TRu practitioners. Prevalence, which corresponds to the number of cases of a disease in a population at a given time, encompassing both new and old cases, would enable us to assess the relevance or otherwise of conducting further, more in-depth studies on the subject. Investigators would also like to clarify the circumstances and factors associated with the injury, in order to establish a true picture of this pathology in France.

Issues In summary, the number of runners is constantly increasing, and TRu seems to be a high-risk activity for the ankle joint. Ankle sprains can lead to significant health consequences, as in the case of chronic ankle instability.

However, there are no studies on the prevalence of chronic ankle instability in trail running. The aim of this study is, therefore, to take stock of chronic ankle instability in trail running in France.

ELIGIBILITY:
Inclusion Criteria:

* Trail Running
* Ultra Trail Running runners
* Having participated́ in at least one Trail Running or Ultra Trail Running competition in their lifetime.
* Over 18 years of age (adult participants)

Exclusion Criteria:

* Adults protected under Article L1121-8 of the French Public Health Code
* Minors
* Adults unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Trail Running racers who have participated in at least one Trail Running competition in their lifetime. Subjects will be recruited via an online questionnaire distributed through various French Trail Running organizations and social networks.
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of chronic ankle instability in trailers | Time 0
  Number of cases among all respondents with a Cumberland Ankle Instability Tool Score ≤ 23 points for the French version end ≤ 25 points for the English version. (validated questionnaire)

SECONDARY OUTCOMES:
Socio-demographic data (1/4) | Time 0
  Average ages among the 3 study populations (in years)
Socio-demographic data (2/4) | Time 0
  Proportion of sex ratios among 3 study populations
Socio-demographic data (3/4) | Time 0
  Proportion of majority training grounds among 3 study populations
Socio-demographic data (4/4) | Time 0
  Proportion of practice statuses among the 3 study populations
Trail running and prevalence reports (1/11) | Time 0
  Proportion of training club members among the 3 populations studied
Trail running and prevalence reports (2/11) | Time 0
  Average years of practice among the 3 populations studied (in years)
Trail running and prevalence reports (3/11) | Time 0
  Average training hours per week among the 3 populations studied (in hours)
Trail running and prevalence reports (4/11) | Time 0
  Average distances covered in training per week among the 3 populations studied (in kilometers)
Trail running and prevalence reports (5/11) | Time 0
  Proportion of competitions per year among the 3 populations studied
Trail running and prevalence reports (6/11) | Time 0
  Average distances covered in competition among the 3 study populations (in kilometers)
Trail running and prevalence reports (7/11) | Time 0
  Average times spent in competition among the 3 populations studied (in hours)
Trail running and prevalence reports (8/11) | Time 0
  Proportions of sprain occurrence times during annual programming among Copers and ICC populations
Trail running and prevalence reports (9/11) | Time 0
  Proportion of sprain occurrence times during sessions among Copers and ICC populations
Trail running and prevalence reports (10/11) | Time 0
  Proportions of sprain occurrence times according to pitch inclination variability in the Copers and ICC populations.
Trail running and prevalence reports (11/11) | Time 0
  Proportion of sprain occurrence times according to variability of terrain characteristics in the Copers and ICC populations.
Associated pathologies (1/2) | Time 0
  Proportions of the presence or absence of musculoskeletal disorders recorded over the past 12 months among the 3 populations studied.
Associated pathologies (2/2) | Time 0
  Proportions and body chart of pathologies among participants having recorded a musculoskeletal disorder in the last 12 months within the 3 populations studied
Medical care (1/3) | Time 0
  Proportion of participants having had or using physiotherapy in the Copers and ICC populations.
Medical care (2/3) | Time 0
  Proportions of medical devices used among Copers and ICC populations
Medical care (3/3) | Time 0
  Proportion of different sprain-related impacts among Copers and ICC populations

CONTACTS AND LOCATIONS:
Overall Officials: Leo Druart, PhD, Principal Investigator — University Grenoble Alpes
Locations (1):
- University Grenoble Alpes, Grenoble, France